CLINICAL TRIAL: NCT06600542
Title: Inari VISION Registry
Status: Recruiting | Type: Observational
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-003
Record Dates: First submitted 2024-08-15; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Inari Medical Commercially Available Devices — Commercially approved Inari Medical devices

SUMMARY:
This registry is a global prospective, non-randomized, multicenter, observational, active post-market data collection of Inari Medical devices and products.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent per institution and geographical requirements
2. Has received treatment with an eligible Inari Medical device. NOTE: If patients are consented prior to their procedure and the procedure does not take place, the patient will be considered a screen failure.
3. Currently within enrollment window relative to their procedure
4. Age ≥ 18 years

Exclusion Criteria:

1. Is or will be inaccessible for registry follow-up
2. Meets exclusion criteria required by local requirements
3. Current or planned participation in another drug or device study that, in the investigator's opinion, would interfere with participation in this registry
4. Is pregnant or breastfeeding at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated with an Inari Medical device.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of device-related, procedure-related, or fatal Adverse Events | Up to 180 days

CONTACTS AND LOCATIONS:
Locations (8):
- Santa Marta, Lisbon, Portugal
- United Kingdom (7):
  - Southmead Hospital Bristol, Bristol
  - Queen Elizabeth University Hospital, Glasgow
  - Northwick Park Hospital, London
  - Royal Free Hospital, London
  - Royal London, London
  - UCLH University College London Hospital, London
  - Royal Victoria Infirmary, Newcastle